CLINICAL TRIAL: NCT02426255
Title: Prospective Cohort of Severe Trauma Patients Hospitalized in West French Intensive Care Units
Brief Title: Post Traumatic Critical Complications: a Prospective Cohort Study (ATLANREA)
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0207 cohorte fiche 2
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Severe Trauma (With or Without Traumatic Brain Injury)
Keywords: Severe trauma; traumatic Brain injury; Hemorrhage
MeSH Terms: conditions — Wounds and Injuries; Brain Injuries, Traumatic; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, sera, peripheral blood mononuclear cells, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: Patients with severe trauma (with or without brain injury) or Patients with hemorrhagic shock Data concerning the ICU stay will be collected for these patients
  Interventions: Other: Collection of medical data from ICU patients

INTERVENTIONS:
Other: Collection of medical data from ICU patients — A code will be applied to each patient included. Medical data such as demography, Simplified Acute Physiological Score II (SAPS II), Sequential Organ Failure Assessment (SOFA), procedures and complications during ICU stay will be collected.

SUMMARY:
The purpose of this observational epidemiological study is to investigate the management and the complications associated with severe trauma. Data will be analysed to answer pre-defined scientific projects and to improve management of these conditions.

DETAILED DESCRIPTION:
Pseudonymized data will be collected by study coordinators in a secured e-database.

Cross audit will be performed to check data.

ELIGIBILITY:
Inclusion Criteria:

* severe trauma
* and/or traumatic brain injury
* and/or hemorrhage

Exclusion Criteria:

* Consent withdrawal

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in ICU for severe trauma
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-03-29 (Actual); Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
in ICU stay complications | Within the 28 first days after ICU admission date
  Nosocomial Infections (epidemiology, risk factors, antibiotic susceptibility of pathogens) Organ failures (incidence, risk factors) Bleeding, hemorrhage Intra-cranial hypertension, brain ischemia Mechanical ventilation weaning, extubation failure

SECONDARY OUTCOMES:
Duration of mechanical ventilation | in ICU (up to 90 days)
ICU length of stay | in ICU (up to 90 days)

OTHER OUTCOMES:
Death | in ICU (up to 90 days)

CONTACTS AND LOCATIONS:
Overall Officials: Karim ASEHNOUNE, PhD, MD, Study Chair
Locations (5):
- France (5):
  - Angers University Hospital, Angers
  - Nantes University Hospital, Nantes
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours